CLINICAL TRIAL: NCT07203196
Title: Circadian Health Regulation and Optimization for Rejuvenation Outcomes: The CHRONO Study
Brief Title: Circadian Health Regulation and Optimization for Rejuvenation Outcomes
Acronym: CHRONO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Salk Institute for Biological Studies (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Satchidananda Panda, PhD, Professor, Salk Institute for Biological Studies
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 812811
Record Dates: First submitted 2025-09-12; First posted 2025-10-02 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Aging, Healthy; Blood Sugar; High; Blood Sugar (Glucose) Control; Time Restricted Eating; Circadian Dysregulation
Keywords: Time restricted eating; healthy aging; circadian disruption
MeSH Terms: conditions — Hyperglycemia; Intermittent Fasting; Chronobiology Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Circadian Rhythm Optimization (Experimental): Each participant will be provided with a personalized plan centered on synchronizing their behavior with their endogenous rhythm.
  Interventions: Behavioral: Circadian Rhythm Optimization

INTERVENTIONS:
Behavioral: Circadian Rhythm Optimization — Participants will follow a Mediterranean diet while consuming all calories within a personalized 8-10 hour daytime window. They will increase daytime light exposure to at least one hour per day, engage in a minimum of 150 minutes of moderate-intensity aerobic exercise each week (including at least two sessions lasting no less than 60 minutes), maintain a consistent 7-9 hour sleep schedule, and take supplements as recommended based on individual needs. Participants will also record all food and beverage intake, as well as exercise, using the myCircadianClock app.

SUMMARY:
In this single arm intervention trial, the investigators will assess the impact of a personalized lifestyle plan, centered on supporting biological rhythms, on blood sugar levels, physical, cognitive and immune function in older adults with a habitual eating window of 12 hours or more, and elevated blood glucose levels.

All participants will be provided with a personalized circadian rhythm optimization plan (CRO) centered on improving (1) diet, (2) exercise (3) sleep habits based on their body's natural rhythms. The study includes a 2-week screening/baseline assessments, with follow-up health assessments at 2-months.

DETAILED DESCRIPTION:
The purpose of this study is to assess if modifying lifestyle behaviors such as improving nutrition quality while consolidating caloric intake to a consistent 8-10 hour window, incorporating regular exercise and ensuring a consistent sleep window will help improve glucose (sugar) regulation, physical, cognitive and immune function and improve other markers of metabolic, cardiovascular health and aging (i.e. lipid levels, inflammation markers, etc.).

Circadian clocks ("circa" means approximately and "dia" means day) are daily rhythms in physiology and behavior (activity, sleep, eating pattern) that help the body anticipate and adapt to predictable events in the environment. These rhythms are generated and maintained by biological clocks that are present in the brain and almost every organ. Remarkably, even in the absence of any timing information from a device, the human body can keep track of time and thereby help us eat and sleep at optimum times. However, our lifestyle and work schedules can lead us to eat, exercise, and sleep at times that the clocks in our body are not prepared for. When these abnormal daily patterns continue for several weeks or years, it can affect our health in many ways including increased body weight, poor sleep, and elevated risk for various chronic diseases.

A growing body of preclinical research has shown that synchronizing behaviors, such as food intake, exercise, and light exposure, with the body's biological clock improves skeletal muscle function, cognitive performance, and inflammatory markers. Clinical studies have further validated these findings, showing that circadian-based interventions, such as time-restricted eating (TRE), which restricts all caloric intake to a personalized consistent daily eating window, daytime light exposure and exercise have been shown to improve mood, sleep quality and cardiometabolic health. Despite these promising individual findings, no study has comprehensively examined the combined effects of TRE, structured exercise and optimized sleep schedule as an integrated strategy to restore circadian alignment and reverse key physiological markers of aging in older adults.

In this study, the investigators are interested in evaluating the effects of modifying eating, activity and sleeping patterns on age related health outcomes in older adults with elevated blood sugar levels. All participants will be provided with a personalized circadian rhythm optimization (CRO) program centered on (1) consuming a Mediterranean diet within a personalized 8-10-hour daytime window, (2) increasing daytime light exposure and reducing bright light at night, (3) incorporating 150 minutes of moderate-intensity aerobic exercise each week (4) holding a consistent 7-9 hour sleep schedule (5) taking supplements based on individual needs.

The study is 90-days including a 2-week screening/baseline assessment followed by a 2-week period to developed their personalized plan based off their baseline assessments and finally a 8-week guided intervention period. Health assessments will be taken at screening/baseline, and at 90 days. Assessments will include cognitive function (cognitive assessment battery), physical function (VO2 Max, isometric strength, short physical performance battery), dietary recall (ASA24), blood tests (biomarkers of cardiometabolic health and immune parameters), glycemic regulation (Continuous Glucose Monitors), body composition ( bioelectrical impedance scan), dietary intake (logged on the myCircadianClock smartphone app), sleep and quality of life questionnaires, and activity, sleep, and wrist temperature (actigraphy watch) and subclavian and ankle surface temperature (non-invasive temperature sensor).

ELIGIBILITY:
Inclusion Criteria:

1. Age: 50-80 years
2. Fasting glucose ≥ 100 mg/dL or HbA1c > 5.6%
3. Own a smartphone (Apple iOS or Android OS)
4. Proficient in reading and speaking in English
5. An eating window ≥12 hour/day
6. Willing to travel to sports facilities for exercise training sessions
7. Participants on cardiovascular medications (HMG CoA reductase inhibitors (statins), metformin, SLGT2 inhibitors, GLP1 receptor agonists other lipid-modifying drugs (including over-the counter drugs such as red yeast rice and fish oil), anti-hypertensive, drugs), are allowed if on a stable dose for 6-months, but dose adjustments are not allowed during the study

Exclusion Criteria:

1. Insufficient dietary logging on the mCC app during screening, defined as less than 7 of 14 days of baseline of dietary logging with a minimum of 2 items a day, at least 5 hours apart
2. Type 1 Diabetes or Insulin-dependent Type 2 Diabetes
3. HbA1C > 9.0%
4. Use of sulfonylurea or insulin within the last 3 months (due to unknown safety with TRE)
5. Change in medications that could impact study outcomes within the past 6 months
6. Change in weight of >4kg in the past 3 months
7. Systolic BP greater than 160 mmHg and/or diastolic BP greater than 110 mmHg at rest
8. Fasting LDL cholesterol greater than 250 mg/dL
9. Fasting triglycerides greater than 500g/dL
10. Variable work hours, such as working night shifts
11. Caregiver for a dependent requiring frequent nocturnal care/sleep interruptions
12. Active tobacco use, illicit drug use, or history of treatment for alcohol abuse in the past 5 years.
13. Travel involving a time zone change of more than 3 hours twice or more during the study period
14. Active treatment for inflammatory and/or rheumatologic disease
15. History of a major adverse cardiovascular event within the past year (acute coronary syndrome, percutaneous coronary intervention, coronary artery bypass graft surgery, hospitalization for congestive heart failure, stroke/transient ischemic attack)
16. Uncontrolled arrhythmia (i.e. rate-controlled atrial fibrillation/atrial flutter are acceptable)
17. Previously diagnosed with sever aortic stenosis
18. Previously diagnosed with sever COPD (FEV1/FVC ratio <.7 & FEV1 (%predicted) <49
19. Orthopedic impairments severely compromising exercise performance
20. BMI <18.5 kg/m2
21. History of thyroid disease requiring dose titration of thyroid replacement medication(s) within the past 6 months (i.e. hypothyroidism on a stable dose of thyroid replacement therapy is not an exclusion).
22. History of adrenal disease in the past 5 years
23. History of malignancy undergoing active treatment, except non-melanoma skin cancer, in the past 5 years
24. History of an eating disorder in the past 5 years
25. History of cirrhosis in the past 5 years
26. History of stage 4 or 5 chronic kidney disease or dialysis in the past 5 years
27. History of HIV/AIDs
28. Currently enrolled in weight-loss or weight-management program
29. Regularly engages in 100 minutes or more of structured exercise
30. VO2 max threshold is above average for that individuals age group [78]
31. Uncontrolled psychiatric disorder including prior hospitalization

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
HbA1c (%) | Baseline and 90 days
  HbA1c levels (%) as assessed by fasting blood draw

SECONDARY OUTCOMES:
Grip Strength | Baseline and 90 days
  Maximal grip force (Kg)
Isometric Knee Strength | Baseline and 90 days
  Maximal force output for knee flexion and extension (Kg)
VO2 Max | Baseline and 90 days
  Maximal oxygen consumption (mL/kg/min).
Time to 85% of Age Predicted Maximal Heart Rate | Baseline and 90 days
  Time to 85% of age predicted maximal heart rate (mins).
Flanker Inhibitory and Control and Attention Test (Fully-Corrected T-score) | Baseline and 90 days
  Flanker Inhibitory and Control and Attention Test (Fully-Corrected T-score) assessed through NIH cognitive assessment battery. The score compares an individual's cognitive performance to a nationally representative norming sample correcting for age, sex, race/ethnicity, and educational attainment.
Dimensional Change Card Sort (Fully-Corrected T-score) | Baseline and 90 days
  Dimensional Change Card Sort (Fully-Corrected T-score) assessed through NIH cognitive assessment battery. The score compares an individual's cognitive performance to a nationally representative norming sample correcting for age, sex, race/ethnicity, and educational attainment.
Pattern Comparison Processing Speed Test (Fully-Corrected T-score) | Baseline and 90 days
  Pattern Comparison Processing Speed Test (Fully-Corrected T-score) assessed through NIH cognitive assessment battery. The score compares an individual's cognitive performance to a nationally representative norming sample correcting for age, sex, race/ethnicity, and educational attainment.
Picture Sequence Memory test (Fully-Corrected T-score) | Baseline and 90 days
  Picture Sequence Memory test (Fully-Corrected T-score) assessed through NIH cognitive assessment battery. The score compares an individual's cognitive performance to a nationally representative norming sample correcting for age, sex, race/ethnicity, and educational attainment.
Trail Making Test | Baseline and 90 days
  Trail making test part A and B will be assessed by the time to completion (seconds) for each assessment.
Glucagon (pg/mL) | Baseline and 90 days
  Glucagon (pg/mL) assessed through fasting blood draw
Leptin (ng/mL) | Baseline and 90 days
  Leptin (ng/mL) assessed through fasting blood draw
IL-1α (pg/mL) | Baseline and 90 days
  IL-1α (pg/mL) assessed through fasting blood draw
IL-1β (pg/mL) | Baseline and 90 days
  IL-1β (pg/mL)assessed through fasting blood draw
IL-2 (pg/mL) | Baseline and 90 days
  IL-2 (pg/mL) assessed through fasting blood draw
IL-3 (pg/mL) | Baseline and 90 days
  IL-3 (pg/mL) assessed through fasting blood draw
IL-4 (pg/mL) | Baseline and 90 days
  IL-4 (pg/mL) assessed through fasting blood draw
IL-5 (pg/mL) | Baseline and 90 days
  IL-5 (pg/mL) assessed through fasting blood draw
IL-6 (pg/mL) | Baseline and 90 days
  IL-6 (pg/mL) assessed through fasting blood draw
IL-7 (pg/mL) | Baseline and 90 days
  IL-7 (pg/mL) assessed through fasting blood draw
IL-8 | Baseline and 90 days
  IL-8 (pg/mL) assessed through fasting blood draw
IL-9 (pg/mL) | Baseline and 90 days
  IL-9 (pg/mL) assessed through fasting blood draw
IL-10 (pg/mL) | Baseline and 90 days
  IL-10 (pg/mL) assessed through fasting blood draw
IL-12p70 (pg/mL) | Baseline and 90 days
  IL-12p70 (pg/mL) assessed through fasting blood draw
IL-13 (pg/mL) | Baseline and 90 days
  IL-13 (pg/mL) assessed through fasting blood draw
IL-15 (pg/mL) | Baseline and 90 days
  IL-15 (pg/mL) assessed through fasting blood draw
IL-16 (pg/mL) | Baseline and 90 days
  IL-16 (pg/mL) assessed through fasting blood draw
IL-17A (pg/mL) | Baseline and 90 days
  IL-17A (pg/mL) assessed through fasting blood draw
IL-17F (pg/mL) | Baseline and 90 days
  IL-17F (pg/mL) assessed through fasting blood draw
IL-18 (pg/mL) | Baseline and 90-days
  IL-18 (pg/mL) assessed through fasting blood draw
IL-20 (pg/mL) | Baseline and 90 days
  IL-20 (pg/mL) assessed through fasting blood draw
IL-21 (pg/mL) | Baseline and 90 days
  IL-21 (pg/mL) assessed through fasting blood draw
IL-22 (pg/mL) | Baseline and 90 days
  IL-22 (pg/mL) assessed through fasting blood draw
IL-23 (pg/mL) | Baseline and 90 days
  IL-23 (pg/mL) assessed through fasting blood draw
IL-27 (pg/mL) | Baseline and 90 days
  IL-27 (pg/mL) assessed through fasting blood draw
IL-28 (pg/mL) | Baseline and 90 days
  IL-28 (pg/mL) assessed through fasting blood draw
IL-33 (pg/mL) | Baseline and 90 days
  IL-33 (pg/mL) assessed through fasting blood draw
MCP-1 (pg/mL) | Baseline and 90 days
  MCP-1 (pg/mL) assessed through fasting blood draw
MCP-2 | Baseline and 90 days
  MCP-2 (pg/mL) assessed through fasting blood draw
MCP-3 (pg/mL) | Baseline and 90 days
  MCP-3 (pg/mL) assessed through fasting blood draw
MCP-4 (pg/mL) | Baseline and 90 days
  MCP-4 (pg/mL) assessed through fasting blood draw
TGFα (pg/mL) | Baseline and 90 days
  TGFα (pg/mL) assessed through fasting blood draw
TNFβ (pg/mL) | Baseline and 90 days
  TNFβ (pg/mL) assessed through fasting blood draw
EGF (pg/mL) | Baseline and 90 days
  EGF (pg/mL) assessed through fasting blood draw
TNF-α (pg/mL) | Baseline and 90 days
  TNF-α (pg/mL) assessed through fasting blood draw
Ghrelin (pg/mL) | Baseline and 90-days
  Ghrelin (pg/mL) assessed through fasting blood draw
IGF-1 (ng/mL) | Baseline and 90 days
  IGF-1 (ng/mL) assessed through fasting blood draw
IGF-2 (ng/mL) | Baseline and 90 days
  IGF-2 (ng/mL) assessed through fasting blood draw
IL-1RA (pg/mL) | Baseline and 90 days
  IL-1RA (pg/mL) assessed through fasting blood draw
TRAIL (pg/mL) | Baseline and 90 days
  TRAIL (pg/mL) assessed through fasting blood draw
VEGF-A (pg/mL) | Baseline and 90 days
  VEGF-A (pg/mL) assessed through fasting blood draw
IGFBP-1 (ug/mL) | Baseline and 90 days
  IGFBP-1 (ug/mL) assessed through fasting blood draw
GIP (pg/mL) | Baseline and 90-days
  GIP(pg/mL) assessed through fasting blood draw
GLP-1 (pmol/L) | Baseline and 90 days
  GLP-1 (pmol/L) assessed through fasting blood draw.
Total Recall (T-score) | Baseline and 90-days
  Total Recall (T-score) as assessed through Hopkins Verbal Learning Test - Revised. T-score is adjusted for participant's age.
Delayed Recall (T-score) | Baseline and 90-days
  Delayed Recall (T-score) as assessed through Hopkins Verbal Learning Test. T-score is adjusted for participant's age.
Retention Percentage (T-score) | Baseline and 90-days
  Retention Percentage (T-score) as assessed through Hopkins Verbal Learning Test - Revised. T-score is adjusted for participant's age.
Recognition Discrimination Index (T-score) | Baseline and 90-days
  Recognition discrimination index as assessed through Hopkins Verbal Learning Test-Revised. T-score is adjusted for participant's age.
Cognition Fluid Composite (Fully-Corrected T-score) | Baseline and 90-days
  Cognition Fluid Composite (Fully-Corrected T-score) as assessed through a composite score of several tests, namely the Flanker inhibitory control and attention test, the dimensional change card sort test, the picture sequence memory test, the list sorting working memory test, and the pattern comparison processing speed test. The score compares an individual's cognitive performance to a nationally representative norming sample correcting for age, sex, race/ethnicity, and educational attainment.

OTHER OUTCOMES:
Total Body Fat Mass (kg) | Baseline and 90 days
  Total Body Fat Mass (kg) assessed by bioelectrical impedance scan
Fat Free Mass | Baseline and 90 days
  Whole body fat free mass (kg) assessed by bioelectrical impedance scan
Intra-Daily Glycemic Variability: CONGA (A.U.) | Baseline and 90-days
  Continuous Overall Net Glycemic Action (CONGA) assessed via continuous glucose monitor
Inter-Daily Glycemic Variability: MODD (mg/dL) | Baseline and 90 days
  Mean of Daily Differences (MODD) assessed via continuous glucose monitor
Glycemic Variability: MAGE (mg/dL) | Baseline and 90 days
  Mean Amplitude of Glycemic Excursions (MAGE) assessed by continuous glucose monitor
Mean Glucose (mg/dL) | Baseline and 90 days
  Mean Glucose assessed by continuous glucose monitor
Fasting Glucose | Baseline and 90 days
  Fasting Glucose (mg/dL) assessed through fasting blood draw
Fasting Insulin | Baseline and 90 days
  Fasting insulin (μU/mL) assessed through fasting blood draw
HOMA-IR | Baseline and 90 days
  HOMA-IR assessed through fasting blood draw
Skin Surface Temperature | Baseline and 90 days
  Mean daily Skin surface temperature at the wrist, ankle and subclavian region of the chest (Degrees C) assessed through actigraphy watch and non-invasive skin temperature probe.
Short Physical Performance Battery | Baseline and 90 days
  A sum of the scores from the Chair Stand Test , Gait Speed Test, Side-By-Side- Stand, Semi-Tandem Stand & Tandem Stand Balance Tests. The scoring for each assessment will be based off the previously established and widely used Short Physical Performance Battery Protocol and score sheet where the Chair Stand Test , Gait Speed Test and balance tests scoring are based off the participants ability to rise from the chair, duration is takes to cover 4m distance (seconds) and duration they are able to balance (seconds) respectively.
Quality of Life Assessment | Baseline and 90 days
  Short-Form 36 (SF-36) Survey. Scores range from 0-100 (an average of all questions which each have a 0-100 scale), with 100 indicating better physical and emotional health.
Triglycerides (mg/dL) | Baseline and 90 days
  Triglycerides (mg/dL) from fasted blood draw.
Total Cholesterol (mg/dL) | Baseline and 90 days
  Total cholesterol (mg/dL) from fasted blood draw.
HDL-cholesterol (mg/dL) | Baseline and 90 days
  HDL-cholesterol (mg/dL) from fasted blood draw.
hs-CRP (mg/dL) | Baseline and 90 days
  hs-CRP (mg/dL) from a fasted blood draw.
LDL Particle number (nmol/L) | Baseline and 90 days
  LDL Particle number (nmol/L) assessed by NMR lipoprotein profiles from a fasted blood draw.
Apo A (mg/dL) | Baseline and 90 days
  Apo A (mg/dL) assessed by NMR lipoprotein profiles from a fasted blood draw.
Apo B (mg/dL) | Baseline and 90 days
  Apo B (mg/dL) assessed by NMR lipoprotein profiles from a fasted blood draw.
Apo A/B ratio | Baseline and 90 days
  Apo A/B ratio assessed by NMR lipoprotein profiles from a fasted blood draw.
Very Low Density Lipoprotein (VLDL) Size (nm) | Baseline and 90 days
  VLDL size (nm) assessed by NMR lipoprotein profiles from a fasted blood draw.
HDL Particle number (umol/L) | Baseline and 90 days
  HDL Particle number (umol/L) assessed by NMR lipoprotein profiles from a fasted blood draw.
Thyroid-Stimulating Hormone (µU/mL) | Baseline and 90 days
  Thyroid-Stimulating Hormone (µU/mL) assessed through fasting blood draw
Sex Hormone Binding Globulin (nmol/L) | Baseline and 90 days
  Sex Hormone Binding Globulin (nmol/L) assessed through fasting blood draw
Gamma-Glutamyl Transferase (IU/L) | Baseline and 90 days
  Gamma-Glutamyl Transferase (IU/L) assessed through fasting blood draw
Cystatin C (mg/L) | Baseline and 90 days
  Cystatin C (mg/L) assessed through fasting blood draw
N-terminal pro-B-type natriuretic peptide (pg/mL) | Baseline and 90 days
  N-terminal pro-B-type natriuretic peptide (pg/mL) assessed through fasting blood draw
Vitamin D | Baseline and 90-days
  Vitamin D levels (ng/mL) assessed through fasting blood draw.

CONTACTS AND LOCATIONS:
Overall Officials: Satchidananda Panda, PhD, Principal Investigator — Salk Institute for Biological Studies; Pam Taub, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators will report deidentified individual participant data for outcomes that are reported in scientific publications (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available within 1 month of publication with no set end date (minimum of 5 years).
Access Criteria: Data will be available to anyone who wants to access it through a data depository that will be disclosed at the time of publication.